CLINICAL TRIAL: NCT06350032
Title: Open-label, Single-arm, Non-controlled Trial to Evaluate Safety and Tolerability of Treprostinil Sodium in Children Below the Age of 18 Years Diagnosed With Pulmonary Arterial Hypertension (PAH)
Brief Title: Investigational Trial to Evaluate Safety and Tolerability of Treprostinil in Children Diagnosed With PAH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREPaed; 2023-505082-91-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-19; First posted 2024-04-05 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- preservative-free parenteral treprostinil (Experimental): Patients will be treated with either SC or IV preservative-free treprostinil formulation. Dosing is not stipulated by the study protocol and will be done according to investigators discretion based on patient needs.
  Interventions: Drug: preservative-free parenteral treprostinil

INTERVENTIONS:
Drug: preservative-free parenteral treprostinil — Continuous infusion of either SC or IV preservative-free treprostinil. The dosing is not stipulated by the study protocol and will be done according to patient needs.

SUMMARY:
The goal of this clinical trial is to evaluate safety and tolerability of preservative-free parenteral treprostinil in paediatric patients with PAH (PH Group 1) who are below 18 years of age. The main question it aims to answer is:

• if preservative-free parenteral treprostinil is safe and tolerable in the treatment of paediatric PAH in patients who are either prostacyclin-naïve or have been previously treated with commercially available parenteral treprostinil formulations.

Participants will receive either subcutaneous (SC) or intravenous (IV) preservative-free treprostinil and will be observed for 5 months (20 weeks ± 1 week).

DETAILED DESCRIPTION:
In this study, a preservative-free treprostinil solution provided in a single-use vial will be used. Efficacy of treprostinil for the treatment of PAH in pulmonary hypertension (PH) Group 1 in children is reported throughout literature. However, since the removal of the preservative might impact the safe use of the parenteral solution for infusion, the safety profile of the newly developed preservative-free treprostinil solution will be assessed within this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the parents or the legal representatives and written assent from appropriately aged participants
2. Males or females from birth to under 18 years of age at the time informed consent was signed
3. Confirmed diagnosis of severe PAH classified as PH Group 1 requiring a treatment with prostacyclin infusion
4. Current diagnosis of PAH confirmed by right heart catheterisation (RHC) at screening or by historical RHC prior to screening with following haemodynamic findings:

   * Mean pulmonary arterial pressure (mPAP) >20 mmHg
   * Pulmonary vascular resistance Index (PVRI) >3 Wood Units (WU) m² If RHC is not possible due to medical reasons (e.g. neonates and infants), the confirmation by ECHO at the screening is sufficient.
5. Prostacyclin naïve or patients pre-treated with SC or IV treprostinil prior to screening
6. A subject is eligible to participate in this study, as assessed by the investigator, if they are of:

   * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,
   * Child-bearing potential - has a negative pregnancy test and is not lactating and, if sexually active, agrees to continue to use 2 reliable methods of contraception until study completion and for at least 30 days following the last dose of study drug. Examples of reliable birth control methods include true abstinence as a lifestyle choice (periodic sexual abstinence method is not acceptable); the use of oral contraceptives; a reliable barrier method of birth control (diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices)

Exclusion Criteria:

1. Known intolerance to prostacyclin analogues
2. PH related to conditions other than specified above
3. Unrepaired congenital heart disease if surgery is planned within next 5 months
4. Subjects diagnosed with any lung disease
5. Acutely decompensated heart failure within previous 30 days from screening
6. Subjects who have had an atrial septostomy or potts shunt within the previous 6 months of screening
7. Any clinically significant laboratory abnormality that precludes initiation or continuation of treprostinil therapy
8. Moderate to severe hepatic dysfunction as defined by elevated liver function tests (aspartate aminotransferase or alanine aminotransferase) ≥3 times the upper limit of normal at Screening, or Child Pugh class B or C hepatic disease
9. Subjects who are pregnant or breastfeeding
10. Haematological abnormalities (e.g., severe anaemia, Hgb <10 g/dL, leukopenia, White Blood Cells (WBC) <2500/μL)
11. History of substance use disorder, unless a proof of abstinence ≥1 year is provided
12. Other concurrent severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
13. Participation in another clinical trial of an investigational drug or device (including with placebo) within 30 days or 5 half-lives prior to screening, which-ever is longer
14. Patients not able to handle pumps and infusion site if there is no parent, family member, guardian present in their household taking over pump handling or if they are not treated in hospital set-up

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and seriousness of adverse events and adverse drug reactions | 5 months (20 weeks ± 1 weeks)
  The frequency and seriousness of adverse events and adverse drug reactions during the first 5 months (20 weeks ± 1 weeks) of treatment according to Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).

OTHER OUTCOMES:
Change from baseline in quality of Life (QoL) | 5 months (20 weeks ± 1 weeks)
  Change from baseline in quality of Life (QoL) as assessed by the Pediatric Quality of Life Inventory (PedsQoL Version 4.0) questionnaire.
  Rating from 0 (never) to 4 (almost always) per question. Questionnaire will be completed by pediatric patient (version appropriate for age group) and parents/caregivers.
Change from baseline in 6-minute walk distance (6MWD) | 5 months (20 weeks ± 1 weeks)
  Change from baseline in 6MWD (patients > 6 years)
Change from baseline in World Health Organization Functional Class (WHO FC) | 5 months (20 weeks ± 1 weeks)
  Change in WHO FC class assessment based on current PH guidelines ranging from class I to class IV, whereas class IV means severe limitations.
Change from baseline in echocardiography (ECHO) parameters - RA/RV enlargement | 5 months (20 weeks ± 1 weeks)
  right atrium (RA) / right ventricle (RV)
Change from baseline in echocardiography (ECHO) parameters - RV systolic dysfunction | 5 months (20 weeks ± 1 weeks)
Change from baseline in echocardiography (ECHO) parameters - RV/LV end-systolic ratio (PSAX) | 5 months (20 weeks ± 1 weeks)
  RV / left ventricle (LV)
Change from baseline in echocardiography (ECHO) parameters - tricuspid annular plane systolic excursion (TAPSE) | 5 months (20 weeks ± 1 weeks)
Change from baseline in echocardiography (ECHO) parameters - S/D ratio (TR jet) | 5 months (20 weeks ± 1 weeks)
Change from baseline in echocardiography (ECHO) parameters - Pulmonary Artery Acceleration Time (PAAT) | 5 months (20 weeks ± 1 weeks)
Change from baseline in echocardiography (ECHO) parameters - pericardial effusion | 5 months (20 weeks ± 1 weeks)
Change from baseline in echocardiography (ECHO) parameters - eccentricity index | 5 months (20 weeks ± 1 weeks)
Change from baseline in echocardiography (ECHO) parameters - acceleration time | 5 months (20 weeks ± 1 weeks)
Change from baseline in plasma N-terminal pro-brain natriuretic peptide (NT-proBNP) levels | 5 months (20 weeks ± 1 weeks)
Treprostinil plasma concentration | 5 months (20 weeks ± 1 weeks)
  For treprostinil plasma concentration analysis one 0,5 ml blood sample for patients ≤ 20 kg and one 1ml blood (K3-EDTA) sample for patients > 20kg will be taken.

CONTACTS AND LOCATIONS:
Locations (5):
- Medizinische Universität Wien, Vienna, Vienna, Austria
- Necker-Enfants Malades Hospital, Paris, Paris, Paris, France
- Gottsegen National Cardiovascular Center, Budapest, Budapest, Hungary
- Pediatric Cardiac Center, Bratislava, Slovakia
- Ramón y Cajal University Hospital, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No